CLINICAL TRIAL: NCT07335627
Title: Clindamycin as Antimicrobial Treatment for Streptococcus Spp. PeRiprosthetic Infection
Acronym: CASPR
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9536
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Streptococcus Infection
Keywords: Streptococcus Infection; Clindamycin; Antimicrobial Treatment; Osteoarticular infections; Amoxicillin
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clindamycin is an antibiotic with several advantages: high oral bioavailability and good bone and joint penetration. In France, it is a recommended drug for other types of Streptococcus spp. osteoarticular infections and can be used as an alternative to amoxicillin for periprosthetic infections, including when implants are retained.

The hypothesis of this study is that clindamycin is no less effective than other drugs commonly used to treat periprosthetic Streptococcus spp. infections.

The primary objective of this study is to evaluate the success rate of Streptococcus spp. periprosthetic joint infections treated with clindamycin compared to other antibiotic treatments.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (aged 18 years or older) at the time of surgery for infection
* Probable or proven periprosthetic infection with Streptococcus spp. according to EBJIS diagnostic criteria
* Patient operated on in one of the associated centers between 2013 and 2024

Exclusion Criteria:

* Patient who underwent joint resection or amputation
* Patient who was treated with suppressive antibiotic therapy (defined as antibiotic treatment lasting more than 6 months) which was decided upon prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Adult patient at the time of surgery for infection with a probable or proven periprosthetic infection with Streptococcus spp. according to EBJIS diagnostic criteria
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07-21 (Estimated)

PRIMARY OUTCOMES:
Therapeutic success of the medical-surgical strategy | One year after the end of antibiotic treatment
  Therapeutic success of the medical-surgical strategy defined as: patient showing no clinical signs of infection, no need for repeat surgery one year after the end of antibiotic treatment, and no repeat antibiotic treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Orthopédique Septique - CHU de Strasbourg - France, Strasbourg, France